CLINICAL TRIAL: NCT02162004
Title: Sensor-Augmented Continuous Correction in Insulin Pump-Treated Type 1 Diabetes
Brief Title: Continuous Correction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problems
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Signe Schmidt, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC2014
Record Dates: First submitted 2014-06-02; First posted 2014-06-12 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2015-02

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Continuous Glucose Monitoring; Insulin pump; Sensor-augmented pump; Continuous correction of high blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous correction (Experimental): The insulin pump is set to automatically deliver the patient's usual insulin basal rate. The insulin pump bolus calculator is run every 10 minutes by the attending physician. Bolus calculations are based on glucose sensor values.
  Interventions: Procedure: Continuous Correction
- Control (No Intervention): Regular sensor-augmented pump therapy.

INTERVENTIONS:
Procedure: Continuous Correction
  Arms: Continuous correction

SUMMARY:
The potential of currently available diabetes technologies could be further exploited. The investigators propose that sensor-augmented insulin pump therapy may be improved by continuous correction, i.e. continuous evaluation of the need for correction boluses. In practice, this is carried out by running the bolus calculator every 10 minutes. The glucose sensor will provide the bolus calculator with glucose input. Many times, the bolus calculator will come to the result that no insulin is needed. However, when the blood glucose is above the pre-set target value and a correction bolus is needed, an appropriate bolus is automatically delivered by the insulin pump.

The investigators hypothesize that sensor-augmented continuous correction insulin pump therapy can reduce hyperglycemia without increasing the risk of hypoglycemia in patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* T1D ≥ 3 years
* CSII ≥ 1 year
* HbA1c ≤ 8.0% (64 mmol/mol)

Exclusion Criteria:

* Pregnancy or nursing
* Hypoglycemia unawareness
* Gastroparesis
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during or within 30 days prior to the study
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of time CGM values are in the target range 3.9-8.0 mmol/l in the time period 8:00-17:00. | Every 5 min for 9 hours on each study day.
  The primary outcome is difference in the percentage of time CGM values are in the target range 3.9-8.0 mmol/l in the time period 8:00-17:00 on CC-days and Control-days.

SECONDARY OUTCOMES:
Mean CGM glucose value. | Every 5 min for 9 hours on each study day.
Percentage of time when CGM values are < 3.9 mmol/l. | Every 5 min for 9 hours on each study day.
Percentage of time when CGM values are > 8.0 mmol/l. | Every 5 min for 9 hours on each study day.
CGM standard deviation. | Every 5 min for 9 hours on each study day.
Number of hypoglycemic episodes. | Every 5 min for 9 hours on each study day.
Amount of insulin delivered. | Every 30 min for 9 hours on each study day.
Positive Incremental Area Under the Curve | Every 5 min for 9 hours on each study day.

OTHER OUTCOMES:
Mean absolute relative difference. | Every 5 min for 9 hours on each study day.
  CGM accuracy will be evaluated with Hemocue glucose values as reference (mean absolute relative difference).

CONTACTS AND LOCATIONS:
Overall Officials: Signe Schmidt, MD, PhD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark